CLINICAL TRIAL: NCT02298699
Title: Biomarker for Sly Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Sly Disease (MPS VII) (BioSly)
Acronym: BioSly
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BSLY 06-2018
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Developmental Delay; Skeletal Abnormalities; Hepatomegaly; Splenomegaly
Keywords: Sly Disease; Biomarker
MeSH Terms: conditions — Learning Disabilities; Hepatomegaly; Splenomegaly; Mucopolysaccharidosis VII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry 10 ml EDTA blood and a dry blood spot filter card are taken. To proof the correct Sly diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of Sly will be done. The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Sly disease or high-grade suspicion for Sly disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Sly disease from blood (plasma)

DETAILED DESCRIPTION:
Mucopolysaccharidosis type VII (also known as Sly syndrome or Sly disease) is an inherited disease caused by a lack of the enzyme beta-glucuronidase. This enzyme is needed to break down substances in the body called glycosaminoglycans (GAGs). If the enzyme is not present, GAGs cannot be broken down and they build up in the cells and damage them. This causes a wide range of problems such as short stature, skeletal abnormalities, joint stiffness, enlarged spleen and liver, lung infections, heart problems and hernias. Patients usually die within the first year of life, although some survive into their teenage years.

Mucopolysaccharidosis type VII is a life-threatening disease with many patients dying in early childhood. It also debilitating due to the physical and skeletal abnormalities that occur.

Sly syndrome is characterized by coarse facial features, hepatosplenomegaly, protruding sternum and dystosis multiplex. Dystosis multiplex refers to a constellation of skeletal abnormalities and is characterized by an enlarged skull, thickened calvarium, premature closure of lamboid and sagittal sutures, shallow orbits, enlarged J-shaped sella and abnormal spacing of the teeth with dentigerous cysts. There is anterior hypoplasia of the lumbar vertebrae, the long bone diaphyses are enlarged and an irregular appearance of the metaphyses. The epiphyseal centers not well developed, the pelvis is poorly formed with small femoral heads and coxa valga. The clavicles are short, thick and irregular and the ribs are oar shaped. Phalanges are shortened and trapezoidal in shape.

At the time of designation, mucopolysaccharidosis type VII affected approximately 0.001 in 10,000 people in the European Union (EU)*. This is equivalent to a total of around 50 people, and is below the ceiling for orphan designation, which is 5 people in 10,000.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the parents before any study related procedures
* Patients of both genders older than 2 months
* The patient has a diagnosis of Sly disease or a high-grade suspicion for Sly disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

Positive family anamnesis for Sly disease

Developmental delay and/or progressive mental deterioration

Skeletal abnormalities

Hepatomegaly

Splenomegaly

EXCLUSION CRITERIA:

* No Informed consent from the parents before any study related procedures.
* Patients of both genders younger than 2 months
* No diagnosis of Sly disease or no valid criteria for profound suspicion of Sly disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sly disease or high-grade suspicion for Sly disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Sly disease from blood (plasma) | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided